CLINICAL TRIAL: NCT04422353
Title: The Impact of Video Dance Class and Unsupervised Physical Activity on Parkinson's People During the Covid-19 Pandemic: Interventional
Brief Title: Video Dance Class and Unsupervised Physical Activity During Covid-19 Pandemic in People With Parkinson's Disease
Acronym: PTT-Online
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Aline Nogueira Haas (Unknown); Flávia Gomes Martinez (Unknown)
Responsible Party: Principal Investigator, Leonardo A. Peyré-Tartaruga, Adjunct Professor, Federal University of Rio Grande do Sul
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PTT-Parkinson/COVID19; PTT-Parkinson/COVID19 (Registry Identifier: PTT-Parkinson/COVID19)
Record Dates: First submitted 2020-06-07; First posted 2020-06-09 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Parkinson Disease; Parkinson Disease 10
Keywords: Functionality; movement disorders; rehabilitation; depressive symptoms; quality of life; cognition; self-isolation
MeSH Terms: conditions — Parkinson Disease; Parkinson Disease 10; Movement Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- video Dance classes (Experimental): The dance program consists of dance lessons inspired by Forró rhythm and Samba rhythm.
  Classes will be divided into four stages: Joint warm-up and stretching on the chairs; strengthening, balance, and rhythm exercises with the support of the chair; exercises inspired by the samba and forró (Brazilian ballroom dance) basic steps; and Final cool down. The classes will be held through a recorded video that must be played twice a week. Each video class lasts 30 minutes.
  The video Dance classes will happen in the period of self-isolation and social distance during the Covid-19 pandemic.
  Interventions: Other: Video Dance classes
- Unsupervised physical activities (Active Comparator): The unsupervised physical activity programs will happen in the period of self-isolation and social distance during the Covid-19 pandemic. The classes will be held through a recorded video that must be played twice a week. Each video class lasts 30 minutes.
  Interventions: Other: Unsupervised physical activities
- control group (No Intervention): The control group will be people with PD, engaged, before the Covid-19 pandemic, in the Dance, the Nordic Walk and the Aquatic Jogging extension projects at Federal University of Rio Grande do Sul but did not do any type of physical activity during the Covid-19 pandemic.

INTERVENTIONS:
Other: Video Dance classes — The dance program consists of dance lessons inspired by Forró rhythm and Samba rhythm. The classes will be held through a recorded video that must be played twice a week. Each video class lasts 30 minutes.
  Arms: video Dance classes
Other: Unsupervised physical activities — The classes will be held through a recorded video that must be played twice a week. Each video class lasts 30 minutes.
  Arms: Unsupervised physical activities

SUMMARY:
The aim of this study is to analyze the impact of video dance class and unsupervised physical activity on clinical-functional parameters, self-isolation and non-motors symptoms in people with Parkinson's disease during the Covid-19 pandemic.

DETAILED DESCRIPTION:
Experimental Design: an interventional study. Search Location: Exercise Research Laboratory at the School of Physical Education, Physiotherapy and Dance, Federal University of Rio Grande do Sul, and in the Movement Disorders Outpatient Clinic of the Hospital of Clinicals of Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil. Participants: 60 participants from the Dance, the Nordic Walking, and the Aquatic Jogging extension projects at Federal University of Rio Grande do Sul, both sexes, from 50 to 80 years old, diagnosed with idiopathic PD, will be separate in three groups: Video Dance Classes, in the unsupervised physical activity, and in the control group. Interventions: video dance class, unsupervised physical activity, and a control group. The video dance class program will have a frequency of two sessions per week and a duration of 30 minutes for 12 weeks. The unsupervised physical activity receives an unsupervised home exercise program with a frequency of two sessions per week and a duration of 30 minutes for 12 weeks during the Covid-19 pandemic.

The control group will be people with PD, engaged, before the Covid-19 pandemic, in the Dance, the Nordic Walk and the Aquatic Jogging extension projects at Federal University of Rio Grande do Sul but did not do any type of physical activity during the Covid-19 pandemic.

To evaluate the impacts of the activities during the Covid-19 pandemic, evaluations will be performed by telephone after 60 days of social distance and self-isolation. Outcomes: clinical-functional parameters and non-motor parameters. Data Analysis: Data will be described by average values and standard deviation values. The comparisons between groups will be performed using a Generalized Estimating Equations (GEE) analysis, adopting a level of significance (α) of 0.05. Expected Results: Participants who have remained committed with the video dance class or with the unsupervised physical activity during the Covid-19 pandemic expected to be less affected in the analyzed outcomes, especially in Quality of Life, when compared to the control group. In addition, it is expected that the research results could help to future developments in the scientific, technological, economic, social, and environmental fields.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers
* aged over 50 years
* both sexes
* clinical diagnosis of idiopathic PD
* PD staging between 1 and 4 in Hoehn and Yahr Scale (H&Y)
* Peoples with PD engaged, before the Covid-19 pandemic, in the Dance, the Nordic Walk and the Aquatic Jogging extension projects at Federal University of Rio Grande do Sul.

Exclusion Criteria:

* performing recent surgeries, deep brain stimulation (DBS - Deep Brain Stimulations);
* severe heart diseases, uncontrolled hypertension, myocardial infarction within a period of less than one year, being a pacemaker;
* stroke or other associated neurological diseases; insanity;
* prostheses in the lower limbs;
* without ambulation conditions.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Quality of life (QoL) | Change from baseline at 12 weeks.
  The quality of life (QoL) will be measured by the Parkinson's Disease Quality of life (PDQ-8). PDQ-8 is a reduced version of a specific health status questionnaire comprising 39 items, with 8 items. Respondents are requested to affirm one of five ordered response categories according to how often, due to their PD, they have experienced the problem defined by each item. Each item is grouped into eight scales that are scored by expressing summed item scores as a percentage score ranging between 0 and 100 (100¼more health problems).
Depressive symptoms - Geriatric Depression Scale - 15 item | Change from baseline at 12 weeks.
  This outcome will be measure for the Geriatric Depression Scale - 15 item. The scale consists of 15 dichotomous questions in which participants are asked to answer yes or no about how they felt over the past week (for instance, "Do the patient feel that their life is empty?," Do the patient feel that their situation is hopeless?). Scores range from 0 to 15 with higher scores indicating more depressive symptoms.
Physical Activity - International Physical Activity Questionnaires (IPAQ) | Change from baseline at 12 weeks.
  This outcome will be measure for the International Physical Activity Questionnaires (IPAQ). The IPAQ comprises a set of 4 questionnaires. Long (5 activity domains asked independently) and short (4 generic items) versions for use by either telephone or self-administered methods are available. The purpose of the questionnaires is to provide common instruments that can be used to obtain internationally comparable data on health-related physical activity.

SECONDARY OUTCOMES:
Cognitive function - Montreal Cognitive Assessment by telephone | Change from baseline at 12 weeks.
  Montreal Cognitive Assessment (MoCA) is a brief screening tool for mild cognitive impairment. This evaluation accesses different cognitive domains and investigates the individual's abilities in the following areas: attention and concentration, executive functions, memory, language, visuoconstructive skills, conceptualization, calculation, and orientation. The total score of the MoCA is 30 points, with a score of 26, or more, considered normal and less than 26 is considered a cognitive impairment.
Falls - Falls Efficacy Scale - International | Change from baseline at 12 weeks.
  This outcome will be measure for the Falls - Falls Efficacy Scale - International (FES-I). FES-I can be administered as self-completion questionnaires, or administered verbally as part of a research interview or clinical assessment. To calculate the FES-I score when all items are completed, simply add the scores for each item together to give a total that ranges as follows: minimum 16 (no concern about falling) to maximum 64 (severe concern about falling).
Functional lower extremity strength -Five Times Sit to Stand Test | Change from baseline at 12 weeks.
  The Five Times Sit to Stand Test measures one aspect of transfer skill. This test quantifies functional lower extremity strength and identifies movement strategies a people use to complete the transitional movement.

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo A. Peyré-Tartaruga, PhD, Study Director — Federal University of Rio Grande do Sul
Locations (1):
- Universidade Federal do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alberts JL, Linder SM, Penko AL, Lowe MJ, Phillips M. It is not about the bike, it is about the pedaling: forced exercise and Parkinson's disease. Exerc Sport Sci Rev. 2011 Oct;39(4):177-86. doi: 10.1097/JES.0b013e31822cc71a. PMID 21799425
- [Background] Dereli EE, Yaliman A. Comparison of the effects of a physiotherapist-supervised exercise programme and a self-supervised exercise programme on quality of life in patients with Parkinson's disease. Clin Rehabil. 2010 Apr;24(4):352-62. doi: 10.1177/0269215509358933. PMID 20360152
- [Background] Beato RG, Nitrini R, Formigoni AP, Caramelli P. Brazilian version of the Frontal Assessment Battery (FAB): Preliminary data on administration to healthy elderly. Dement Neuropsychol. 2007 Jan-Mar;1(1):59-65. doi: 10.1590/S1980-57642008DN10100010. PMID 29213369
- [Background] Frazzitta G, Balbi P, Maestri R, Bertotti G, Boveri N, Pezzoli G. The beneficial role of intensive exercise on Parkinson disease progression. Am J Phys Med Rehabil. 2013 Jun;92(6):523-32. doi: 10.1097/PHM.0b013e31828cd254. PMID 23552330
- [Background] Hackney ME, Kantorovich S, Levin R, Earhart GM. Effects of tango on functional mobility in Parkinson's disease: a preliminary study. J Neurol Phys Ther. 2007 Dec;31(4):173-9. doi: 10.1097/NPT.0b013e31815ce78b. PMID 18172414
- [Background] Herman T, Giladi N, Gruendlinger L, Hausdorff JM. Six weeks of intensive treadmill training improves gait and quality of life in patients with Parkinson's disease: a pilot study. Arch Phys Med Rehabil. 2007 Sep;88(9):1154-8. doi: 10.1016/j.apmr.2007.05.015. PMID 17826461
- [Background] Hoehn MM, Yahr MD. Parkinsonism: onset, progression and mortality. Neurology. 1967 May;17(5):427-42. doi: 10.1212/wnl.17.5.427. No abstract available. PMID 6067254
- [Background] Morris M, Iansek R, McGinley J, Matyas T, Huxham F. Three-dimensional gait biomechanics in Parkinson's disease: evidence for a centrally mediated amplitude regulation disorder. Mov Disord. 2005 Jan;20(1):40-50. doi: 10.1002/mds.20278. PMID 15390033
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Reuter I, Mehnert S, Leone P, Kaps M, Oechsner M, Engelhardt M. Effects of a flexibility and relaxation programme, walking, and nordic walking on Parkinson's disease. J Aging Res. 2011;2011:232473. doi: 10.4061/2011/232473. Epub 2011 Mar 30. PMID 21603199
- [Background] Shanahan J, Morris ME, Bhriain ON, Saunders J, Clifford AM. Dance for people with Parkinson disease: what is the evidence telling us? Arch Phys Med Rehabil. 2015 Jan;96(1):141-53. doi: 10.1016/j.apmr.2014.08.017. Epub 2014 Sep 16. PMID 25223491
- [Background] Sharp K, Hewitt J. Dance as an intervention for people with Parkinson's disease: a systematic review and meta-analysis. Neurosci Biobehav Rev. 2014 Nov;47:445-56. doi: 10.1016/j.neubiorev.2014.09.009. Epub 2014 Sep 28. PMID 25268548
- [Background] Tuon T, Valvassori SS, Dal Pont GC, Paganini CS, Pozzi BG, Luciano TF, Souza PS, Quevedo J, Souza CT, Pinho RA. Physical training prevents depressive symptoms and a decrease in brain-derived neurotrophic factor in Parkinson's disease. Brain Res Bull. 2014 Sep;108:106-12. doi: 10.1016/j.brainresbull.2014.09.006. Epub 2014 Sep 28. PMID 25264157
- [Background] Zigmond MJ, Smeyne RJ. Exercise: is it a neuroprotective and if so, how does it work? Parkinsonism Relat Disord. 2014 Jan;20 Suppl 1:S123-7. doi: 10.1016/S1353-8020(13)70030-0. PMID 24262162
- [Background] Helmich RC, Bloem BR. The Impact of the COVID-19 Pandemic on Parkinson's Disease: Hidden Sorrows and Emerging Opportunities. J Parkinsons Dis. 2020;10(2):351-354. doi: 10.3233/JPD-202038. No abstract available. PMID 32250324
- [Background] Victorino DB, Guimaraes-Marques M, Nejm M, Scorza FA, Scorza CA. COVID-19 and Parkinson's Disease: Are We Dealing with Short-term Impacts or Something Worse? J Parkinsons Dis. 2020;10(3):899-902. doi: 10.3233/JPD-202073. No abstract available. PMID 32390643
- [Background] Hong J, Kong HJ, Yoon HJ. Web-Based Telepresence Exercise Program for Community-Dwelling Elderly Women With a High Risk of Falling: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2018 May 28;6(5):e132. doi: 10.2196/mhealth.9563. PMID 29807877
- [Result] Monteiro EP, Franzoni LT, Cubillos DM, de Oliveira Fagundes A, Carvalho AR, Oliveira HB, Pantoja PD, Schuch FB, Rieder CR, Martinez FG, Peyre-Tartaruga LA. Effects of Nordic walking training on functional parameters in Parkinson's disease: a randomized controlled clinical trial. Scand J Med Sci Sports. 2017 Mar;27(3):351-358. doi: 10.1111/sms.12652. Epub 2016 Feb 2. PMID 26833853